CLINICAL TRIAL: NCT06376916
Title: Atrial Tachycardia Reduction With Intravenous Use of Magnesium (ATRIUM) Study: Comparing Magnesium 2g Versus 4g Versus Placebo in the Incidence of Treating AFF RVR
Brief Title: Comparing Magnesium 2g Versus 4g Versus Placebo in the Incidence of Treating AFF RVR
Acronym: ATRIUM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00110863
Record Dates: First submitted 2024-04-15; First posted 2024-04-22 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Tachycardia Atrial; Atrial Fibrillation; Atrial Flutter With Rapid Ventricular Response
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Arm One, Magnesium Sulfate 2g (Experimental): Study drug (Magnesium Sulfate 2 gram/50ml 0.9% NaCl)
  Interventions: Drug: Magnesium Sulfate 2 G
- Experimental Arm Two, Magnesium Sulfate 4g (Experimental): Magnesium Sulfate 4g/50ml 0.9% NaCl
  Interventions: Drug: Magnesium Sulfate 4 G
- Control Arm, normal saline (Placebo Comparator): 50ml 0.9% NaCl
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Magnesium Sulfate 2 G — Magnesium Sulfate 2g for the treatment of atrial fibrillation or atrial flutter with rapid ventricular response (AFF RVR)
  Other Names: Magnesium Sulfate 2 gram/50ml 0.9% NaCl
  Arms: Experimental Arm One, Magnesium Sulfate 2g
Drug: Magnesium Sulfate 4 G — Magnesium Sulfate 4g for the treatment of atrial fibrillation or atrial flutter with rapid ventricular response (AFF RVR)
  Other Names: Magnesium Sulfate 4g/50ml 0.9% NaCl
  Arms: Experimental Arm Two, Magnesium Sulfate 4g
Drug: Saline — The control group will receive a bolus of normal saline of the same volume and infused over 15 minutes.
  Other Names: Control (50ml 0.9% NaCl)
  Arms: Control Arm, normal saline

SUMMARY:
The purpose of this prospective, randomized, double-blinded study is to further evaluate the safety and efficacy of varying doses of intravenous magnesium in the treatment of AFF RVR.

DETAILED DESCRIPTION:
Intravenous magnesium has become a commonly utilized agent in the treatment of cardiac arrhythmias as an adjunct therapy to rate and rhythm control medications, such as its use in atrial fibrillation or atrial flutter with rapid ventricular response (AFF RVR). Though its benefit in the treatment of AFF RVR has been well documented, a consensus on the optimal dosing of magnesium has yet to be achieved. Only one randomized, controlled, double-blinded study has investigated the optimal dosing of magnesium.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years or older
* Able to provide informed consent
* Primary diagnosis AFF RVR greater than or equal to 120 bpm
* Diltiazem as rate control agent
* English speaking

Exclusion Criteria:

* Hemodynamically unstable patients (SBP <90, MAP <65)
* Impaired consciousness
* End stage renal disease on hemodialysis or peritoneal dialysis
* Acute heart failure exacerbation based on clinical diagnosis, physician exam, bedside echo, and/or additional imaging
* Patient in AFF RVR that is highly suspected to be a compensatory mechanism for an alternative clinical diagnosis
* Rhythms other than AF, such as sick sinus syndrome or wide-complex ventricular response
* Acute myocardial infarction
* Pregnancy defined as a positive urine HCG (human chorionic gonadotropin)
* Contraindications to magnesium sulfate (including myasthenia gravis)
* Allergy or sensitivity to any study drugs
* Previously enrolled in this trial during a different patient encounter
* Withdrew from study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Ventricular rate control | Within the first 2 hours of intravenous magnesium administration
  Assessing ventricular rate control within the first 2 hours of intravenous magnesium administration as defined as a ventricular rate of < 120 bpm.

SECONDARY OUTCOMES:
Time to achieve goal HR (heart rate) | 2 hours
  Mean change in heart rate and rhythm after the administration of magnesium sulfate as well as after the administration of diltiazem
Rate of conversion | 2 hours after administration of magnesium
  Rate of conversion to normal sinus rhythm (NSR)
Incidence of hypotension | At 1 and 2 hours after magnesium administration
  SBP < 90 mmHg or MAP (mean arterial pressure) < 65
Change in heart rate | up to 24 hours after magnesium infusion
  Mean change in heart rate up to 24 hours after magnesium infusion
Clinical need for rescue medication administration | 2 hours from diltiazem administration
  Dose and route of rescue medications given (magnesium and diltiazem)
Adverse effects | 2 hours from diltiazem administration
  Patient reported adverse effects (e.g.. flushing, headache, nausea, new onset or worsening lightheadedness since beginning the magnesium infusion)

CONTACTS AND LOCATIONS:
Overall Officials: Travis Hase, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Christ Medical Center Emergency Department (ACMC ED), Oak Lawn, Illinois, United States